CLINICAL TRIAL: NCT05860205
Title: A Feasibility and Pilot Study of a Multiple Component Mobile-aid Pain Reduction Intervention to Decrease Myofascial Pain Syndrome
Brief Title: A Multiple Component Mobile-aid Pain Reduction Intervention to Decrease Myofascial Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kailea Manning (Other)
Collaborators: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor-Investigator, Kailea Manning, Research Coordinator, Auburn University
Organization: Auburn University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPS2022
Record Dates: First submitted 2023-04-18; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial Pain Syndrome; Low Back Pain; Myofascial Trigger Points
MeSH Terms: conditions — Myofascial Pain Syndromes; Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Group 1 (no treatment condition) will only receive educational materials through email and a weekly phone call from the Coordinator to reduce dropouts for 12 weeks. Group 2 will receive the new multiple component mobile-aid pain reduction intervention (MCMAPRI) and sham osteopathic manipulative treatment [OMT] for 12 weeks. Group 3 will receive both MCMAPRI and actual OMT for 12 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will not know if they are assigned to the multiple component mobile-aid pain reduction intervention and sham osteopathic manipulation treatment group or the multiple component mobile-aid pain reduction intervention and actual osteopathic manipulation treatment group. Additionally, the outcomes assessors will not know which groups the participants have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment condition (No Intervention): Group 1 (no treatment condition) will only receive educational materials through email and a weekly phone call from Coordinator to reduce dropouts for 12 weeks.
- Multiple component mobile-aid pain reduction intervention + sham osteopathic manipulation treatment (Active Comparator): Group 2 will receive the new intervention and sham osteopathic manipulative treatment for 12 weeks.
  Interventions: Behavioral: Multiple Component Mobile-Aid Pain Reduction Intervention; Other: Sham Osteopathic Manipulation
- Multiple component mobile-aid pain reduction intervention + osteopathic manipulation treatment (Active Comparator): Group 3 will receive both the multiple component mobile-aid pain reduction intervention and actual osteopathic manipulation treatment for 12 weeks.
  Interventions: Behavioral: Multiple Component Mobile-Aid Pain Reduction Intervention; Other: Osteopathic Manipulation Treatment

INTERVENTIONS:
Behavioral: Multiple Component Mobile-Aid Pain Reduction Intervention — 1.Posture training through the wearable device, UPRIGHT GO. The participant wears the device on their neck. The device provides biofeedback to poor posture with vibrations and tracks posture. 2. A daily core muscle training and stretching exercise program including trunk rotation, lumbar rotation, hip flexor stretch, side plank, glute bridge, suitcase carry, and palloff press. 3. Participants will practice stress reduction through breath focus which will help them to concentrate on deep breathing to help them ignore distracting thoughts and sensations. 4. Strategies to improve daily level of activity including wearing a Garmin device that tracks their daily physical activity and reminds them to walk and the use of the communication principle to assist participants in overcoming barriers to physical activity.
  Arms: Multiple component mobile-aid pain reduction intervention + osteopathic manipulation treatment; Multiple component mobile-aid pain reduction intervention + sham osteopathic manipulation treatment
Other: Osteopathic Manipulation Treatment — Osteopathic Manipulation Treatment (OMT) will be conducted by putting pressure on certain muscles in the back and performing OMT exercises on the patient. The physician will treat participants with OMT twice during month 1 and once during month 2 and 3.
  Arms: Multiple component mobile-aid pain reduction intervention + osteopathic manipulation treatment
Other: Sham Osteopathic Manipulation — The sham osteopathic manipulation treatment (OMT) will be performed by the medical team. Hands will be placed on the patient as if the OMT is being performed. The physician will treat participants with sham OMT twice during month 1 and once during month 2 and 3.
  Arms: Multiple component mobile-aid pain reduction intervention + sham osteopathic manipulation treatment

SUMMARY:
The goal of this clinical trial is to pilot test a newly developed multiple component mobile-aid pain reduction intervention (MCMAPRI) and the feasibility of implementing this intervention in adult patients with myofascial pain syndrome of the low back. The main questions it aims to answer are:

* What are the effects of the MCMAPRI intervention on reducing levels of myofascial pain in adult patients with myofascial pain syndrome of the low back?
* What is the feasibility for implementing the MCMAPRI intervention in adult patients with myofascial pain syndrome of the low back?

Participants will be randomly assigned to one of three groups: no treatment group, MCMAPRI intervention + sham osteopathic manipulation treatment, or MCMAPRI intervention +osteopathic manipulation treatment.

* Participants assigned to the no treatment group will only receive educational materials through email and a weekly phone call from the coordinator to reduce dropouts.
* Participants assigned to the multiple component mobile-aid pain reduction intervention+sham osteopathic manipulation treatment group will be asked to engage in posture training through a wearable device (i.e., UPRIGHT GO), a core muscle training and stretching exercise program, stress reduction through breath focus, and in strategies to improve their level of daily activity (i.e., wearing a Garmin device). This group will receive a sham osteopathic manipulation treatment by placing hands on the patient as if osteopathic manipulation treatment is being performed.
* Participants assigned to the MCMAPRI intervention+sham osteopathic manipulation treatment group will be asked to engage in posture training through a wearable device (i.e., UPRIGHT GO), a core muscle training and stretching exercise program, stress reduction through breath focus, and in strategies to improve their level of daily activity (i.e., wearing a Garmin device). This group will receive actual osteopathic manipulation treatment by putting pressure on certain muscles in the back and performing osteopathic manipulation treatment exercises on the patient.

Researchers will compare the no treatment group, multiple component mobile-aid pain reduction intervention+sham osteopathic manipulation treatment group, and multiple component mobile-aid pain reduction intervention+osteopathic manipulation treatment group to see if there are decreased levels of pain, increased physical activity, better posture, and reduced levels of stress.

DETAILED DESCRIPTION:
Design: A three group randomized control trial will be used to pilot test the effect of our newly created multiple component mobile-aid pain reduction intervention (MCMAPRI) on lowering myofascial pain in the low back and for examining the possibility of implementing this intervention in the desired population. The study will consist of a convenience sample of 30 adult patients who currently have myofascial pain of the low back (i.e., tender knots in the low back). This will be a 12-week study with outcomes measured at Week 1 (T1), Week 8 (T2), and Week 14 (T3). Participants will be randomly placed in one of the following three groups after screening and meeting the study criteria. Group 1 (no treatment condition) will only receive educational materials through email and a weekly phone call from Coordinator to reduce dropouts. Group 2 will receive the new intervention and sham osteopathic manipulative treatment [OMT] for 12 weeks. The multiple component mobile-aid pain reduction intervention will include four components: (1) Posture training through the wearable device, UPRIGHT GO which provides biofeedback to poor posture with vibrations and tracks posture; (2) A daily core muscle training and stretching exercise program including trunk rotation, lumbar rotation, hip flexor stretch, side plank, glute bridge, suitcase carry, and the palloff press exercises; (3) Participants will practice stress reduction through breath focus which will help them to concentrate on deep breathing to help them ignore distracting thoughts and sensations; and (4) Strategies to improve daily level of activity including asking the participants to wear a Garmin device that tracks their daily physical activity and the use of the communication principle to assist participants in overcoming barriers to physical activity. For those who receive multiple component mobile-aid pain reduction intervention, initial training will occur right after the pretest and follow-up training will occur at the midpoint of the program. The sham osteopathic manipulation treatment will be performed by our medical team. Hands will be placed on the patient as if the osteopathic manipulation treatment is being performed. The physician will treat participants with sham osteopathic manipulation treatment twice during month 1 and once during month 2 and 3. Group 3 will receive both multiple component mobile-aid pain reduction intervention and actual osteopathic manipulation treatment. osteopathic manipulation treatment will be conducted by putting pressure on certain muscles in the back and performing osteopathic manipulation treatment exercises on the patient. The physician will treat participants with osteopathic manipulation treatment twice during month 1 and once during month 2 and 3.

ELIGIBILITY:
Inclusion Criteria: (1) Myofascial pain syndrome (MPS) of the low back with myofascial trigger points (MTrPs) as specified by Travell and Simons (2) normal neurological examination including manual muscle testing, sensory exam, and deep tendon reflexes, (3) English-speaking, (4) age 18 - 64 and reside in the community, (5) exhibiting low level of physical activity as defined by 150 minutes of moderate-intense physical activity weekly, and (6) exhibiting poor posture.

Exclusion Criteria: (1) malignancy, (2) major psychiatric disorder, such as bipolar disorder and depression, (3) cognitive impairment, (4) systematic pain condition, such as Fibromyalgia, (5) previous surgical procedures in the spine and/or back within six months, (6) pregnancy, (7) body mass index (BMI) of 40 or higher, (8) any health conditions that would prevent performing the testing and intervention procedures, (9) MPS due to pelvic obliquity, scoliosis, anatomical leg length discrepancies, (10) MPS treatment within the last three months or daily use of opioids, or (11) other contraindications that would prevent receiving proposed interventions as identified by study physicians.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Self-report pain Level | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Patients will be asked to report their pain level verbally using a scale from 0-10 where 0 represents no pain and 10 represents the worst pain they have ever felt.
Pain pressure threshold (PPT) | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  PPT will be measured by applying pressure to the trigger points on the patients back using an algometer device. The patient will be instructed to tell as as soon as they feel pain at which point the device is removed and the total pounds of force that were applied will be recorded.
Elasticity of the Myofascial Trigger Point | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The elasticity of myofascial trigger points will be measured through the analysis of ultrasound images taken.
Depth of the Myofascial Trigger Point | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The depth of the myofascial trigger points in the muscle will be measured through the analysis of ultrasound images taken.
Size of the Myofascial Trigger Point | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The size of the myofascial trigger points will be measured through the analysis of ultrasound images taken.

SECONDARY OUTCOMES:
Pain intensity and interference | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Pain intensity and interference will be measured using the Pain Enjoyment and General Activity (PEG) Scale. The minimum score is 0 and the maximum score is 10. A higher score suggests more intense pain and pain interference, however, this measure is used to track participants' pain over the study to determine if the intervention(s) has been effective for decreasing pain.
Physical functioning/quality of life | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Physical functioning/quality of life will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function - Short Form 6b. The minimum score is 6 and the maximum score is 30. A higher score suggests worse physical functioning and quality of life.
Sleep Disturbance | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Sleep disturbance will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 6a. For the Sleep Disturbance Short Form 6a, the minimum score is 6 and the maximum score is 30. A higher score suggests more sleep disturbance.
Sleep duration | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Sleep disturbance will be measured by the National Institutes of Health (NIH) Common Data Elements (CDE) Sleep duration question. When interpreting the single NIH CDE Sleep duration question, a lower duration of sleep suggests more sleep disturbance.
Pain catastrophizing | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Pain catastrophizing will be measured by the Pain Catastrophizing Scale. The minimum score is 0 and the maximum score is 52. A higher score suggests more pain catastrophizing.
Depression | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Depression will be measured using the Patient Health Questionnaire-2 (PHQ-2) to measure depression. The minimum score is 0 and the maximum score is 6 where a higher score indicates higher levels of depression.
Anxiety | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Anxiety will be measured using the Generalized Anxiety Disorder-2 (GAD-2). The minimum score is 0 and the maximum score is 6. A higher score suggests higher levels of anxiety.
Global satisfaction with treatment | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Global satisfaction with treatment will be measured using the Patient Global Impression of Change (PGIC) Scale. This includes one item with a minimum score of 0 and a maximum score of 6. A higher score represents pain worsening from the time of the study.
Substance use | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Screener will be used to measure substance use. Each item is measured on a 4 point scale where 0 represents Daily or Almost Daily and 4 represents Never. Any score other than 0 suggests a positive screen for substance use.
Sit to Stand test (STS) | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The Sit to Stand test (STS) will be used to measure physical function. This test asks participants to stand up and sit down as fast as they can 5 times while the assessor records the time.
Get Up and Go (GUG) | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The Get Up and Go (GUG) test will be used to measure physical function. This test asks the participant to begin from a seated position, walk to a marked point that is 3meters away, turn around and walk back, ending in a seated position while the assessor records the time it takes to complete.
Six-minute walk | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  The six-minute walk test will also be used to measure physical function. This tests asks participants to walk as far as they can in 6 minutes. Participants will walk back and forth along a pre-measured 30 meter stretch. The assessor will record the total length the participant walked when time is up.
Sensor Parameter - Posture | Baseline (Time 1), Change from Baseline at 6 weeks (Time 2), and Change from Baseline at 12 weeks (Time 3)
  Two hour recording session of the participant sitting at a desk, wearing movement sensors, to determine the percentage of poor posture during that recording session.
Sensor Parameter - Uptime | Continuously for 12 weeks
  Poor posture will be measured by "Uptime" using the UPRIGHT GO sensor daily.
Sensor Parameter - Daily Step Count | Continuously for 12 weeks
  Participants' daily step count will be collected from their Garmin device .
Sensor Parameter - Sleep Hours | Continuously for 12 weeks
  Participants' sleep hours will be collected from their Garmin device.
Sensor Parameter - Stress Scores | Continuously for 12 weeks
  Participants' stress scores will be collected from their Garmin device. Devices will provide a stress level between 0 and 100, which correspond to the following scale:0-25: Resting state, 26-50: Low stress, 51-75: Medium stress, 76-100: High stress.

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Feng Tsai, PhD, Principal Investigator — Auburn University; Joseph Edison, DO, Principal Investigator — Edward Via College of Osteopathic Medicine
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Edward Via College of Osteopathic Medicine (VCOM), Auburn, Alabama

REFERENCES:
- [Background] Dua A, Chang KV. Myofascial Pain Syndrome. 2025 Apr 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK499882/ PMID 29763057
- [Background] Skootsky SA, Jaeger B, Oye RK. Prevalence of myofascial pain in general internal medicine practice. West J Med. 1989 Aug;151(2):157-60. PMID 2788962
- [Background] Botwin KP, Patel BC. Electromyographically guided trigger point injections in the cervicothoracic musculature of obese patients: a new and unreported technique. Pain Physician. 2007 Nov;10(6):753-6. PMID 17987097
- [Background] Iglesias-Gonzalez JJ, Munoz-Garcia MT, Rodrigues-de-Souza DP, Alburquerque-Sendin F, Fernandez-de-Las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in patients with chronic nonspecific low back pain. Pain Med. 2013 Dec;14(12):1964-70. doi: 10.1111/pme.12224. Epub 2013 Aug 15. PMID 23947760
- [Background] Lundberg U, Kadefors R, Melin B, Palmerud G, Hassmen P, Engstrom M, Dohns IE. Psychophysiological stress and EMG activity of the trapezius muscle. Int J Behav Med. 1994;1(4):354-70. doi: 10.1207/s15327558ijbm0104_5. PMID 16250795
- [Background] Tsai PF, Wang CH, Zhou Y, Ren J, Jones A, Watts SO, Chou C, Ku WS. A classification algorithm to predict chronic pain using both regression and machine learning - A stepwise approach. Appl Nurs Res. 2021 Dec;62:151504. doi: 10.1016/j.apnr.2021.151504. Epub 2021 Sep 28. PMID 34815000
- [Background] Boissoneault J, Sevel L, Letzen J, Robinson M, Staud R. Biomarkers for Musculoskeletal Pain Conditions: Use of Brain Imaging and Machine Learning. Curr Rheumatol Rep. 2017 Jan;19(1):5. doi: 10.1007/s11926-017-0629-9. PMID 28144827
- [Background] Chu Y, Zhao X, Han J, Su Y. Physiological Signal-Based Method for Measurement of Pain Intensity. Front Neurosci. 2017 May 26;11:279. doi: 10.3389/fnins.2017.00279. eCollection 2017. PMID 28603478
- [Background] Jiang, M. et al. Ultra-short-term analysis of heart rate variability for real-time acute pain monitoring with wearable electronics. IEEE International Conference on Bioinformatics and Biomedicine (BIBM), 1025-1032 (2017).
- [Background] Tavakolian M, Hadid A. Deep binary representation of facial expressions: A novel framework for automatic pain intensity recognition. In2018 25th IEEE International Conference on Image Processing (ICIP) 2018 Oct 7 (pp. 1952-1956). IEEE.
- [Background] Gupta G, Alok M. Effectiveness of plank exercise in low back pain. Int. J. Sci. Res. 2018;9(5).
- [Background] Withall J, Jago R, Fox KR. Why some do but most don't. Barriers and enablers to engaging low-income groups in physical activity programmes: a mixed methods study. BMC Public Health. 2011 Jun 28;11:507. doi: 10.1186/1471-2458-11-507. PMID 21711514
- [Background] Carroll JK, Fiscella K, Epstein RM, Sanders MR, Williams GC. A 5A's communication intervention to promote physical activity in underserved populations. BMC Health Serv Res. 2012 Oct 30;12:374. doi: 10.1186/1472-6963-12-374. PMID 23110376
- [Background] Calatayud J, Escriche-Escuder A, Cruz-Montecinos C, Andersen LL, Perez-Alenda S, Aiguade R, Casana J. Tolerability and Muscle Activity of Core Muscle Exercises in Chronic Low-back Pain. Int J Environ Res Public Health. 2019 Sep 20;16(19):3509. doi: 10.3390/ijerph16193509. PMID 31547140
- [Background] Zaccaro A, Piarulli A, Laurino M, Garbella E, Menicucci D, Neri B, Gemignani A. How Breath-Control Can Change Your Life: A Systematic Review on Psycho-Physiological Correlates of Slow Breathing. Front Hum Neurosci. 2018 Sep 7;12:353. doi: 10.3389/fnhum.2018.00353. eCollection 2018. PMID 30245619
- [Background] Wandner LD, Domenichiello AF, Beierlein J, Pogorzala L, Aquino G, Siddons A, Porter L, Atkinson J; NIH Pain Consortium Institute and Center Representatives. NIH's Helping to End Addiction Long-termSM Initiative (NIH HEAL Initiative) Clinical Pain Management Common Data Element Program. J Pain. 2022 Mar;23(3):370-378. doi: 10.1016/j.jpain.2021.08.005. Epub 2021 Sep 9. PMID 34508905
- [Background] McCarthy EK, Horvat MA, Holtsberg PA, Wisenbaker JM. Repeated chair stands as a measure of lower limb strength in sexagenarian women. J Gerontol A Biol Sci Med Sci. 2004 Nov;59(11):1207-12. doi: 10.1093/gerona/59.11.1207. PMID 15602077
- [Background] Lord SR, Murray SM, Chapman K, Munro B, Tiedemann A. Sit-to-stand performance depends on sensation, speed, balance, and psychological status in addition to strength in older people. J Gerontol A Biol Sci Med Sci. 2002 Aug;57(8):M539-43. doi: 10.1093/gerona/57.8.m539. PMID 12145369
- [Background] Piva SR, Fitzgerald GK, Irrgang JJ, Bouzubar F, Starz TW. Get up and go test in patients with knee osteoarthritis. Arch Phys Med Rehabil. 2004 Feb;85(2):284-9. doi: 10.1016/j.apmr.2003.05.001. PMID 14966715
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180